CLINICAL TRIAL: NCT04219644
Title: Evaluation and Validation of the "Breatheasy" Respiratory Rate Monitor in Pre-hospital Care
Brief Title: Evaluation of the "Breatheasy" in Pre-hospital Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCH-15-048
Record Dates: First submitted 2018-06-15; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Respiratory

ARMS (1):
- Breathing test or sleep study (Other): To evaluate the usability of the device in non-clinical and clinical settings
  Interventions: Device: Breatheasy device

INTERVENTIONS:
Device: Breatheasy device

SUMMARY:
In the emergency department, a sick child is usually seen first by the nursing staff. Their job is to quickly assess how sick the child is and what immediate care is needed. The nurse will usually use suitable devices to check vital signs, such as body temperature, pulse rate and blood oxygen levels. However, normally the respiratory rate has to be manually counted (this is the average number of breaths taken each minute) because there is no suitable device which can automatically do this assessment. To overcome this problem we have produced a noncontact device that can automatically measure respiratory rate in children. The device has been designed using the latest technology and works by directly sensing the air coming from the nose or the mouth when held at about 20 cm from the face. It has been tested on adults and children and compared to the usual methods of measuring respiratory rate. We have used comments and Suggestions from members of the public and healthcare professionals from hospital, general practice and the ambulance service to help us develop the device. With this study, we explore the applicability and usefulness of the device in a range of difference clinical and nonclinical settings. Its performance will be carefully evaluated on children and adults in children's nurseries, schools, university, hospital emergency departments, general practice surgeries and ambulances. In the future, when using the device nursing staff will easily be able to measure each child's respiratory rate so that the most seriously ill children will be identified earlier and get correct treatment more quickly. This will ensure that the right children get admitted to intensive care units sooner and, in some cases, deaths will be prevented.

ELIGIBILITY:
Inclusion Criteria:

- Any adult or child within each setting, of any age with any clinical condition, as this will reflect clinical practice.

Exclusion Criteria:

* Patients deemed too unwell to consent to the procedures or requiring emergency treatment will not be approached.
* For the purposes of this feasibility study, families whose first language is not English will be excluded, to save translation and interpretation costs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Respiratory rate using the prototype device | 5 minutes
  In the future, when using the device nursing staff will easily be able to measure each child's respiratory rate so that the most seriously ill children will be identified earlier and get correct treatment more quickly.